CLINICAL TRIAL: NCT05670912
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center II Clinical Trial to Evaluate the Efficacy and Safety of Wei Li Bai Capsules in the Treatment of Mild to Moderate Alzheimer's Disease
Brief Title: Efficacy and Safety of Wei Li Bai Capsules in the Treatment of Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the inability to complete subject enrollment and follow-up as originally scheduled, coupled with funding shortages and overall strategic adjustments from the sponsor, the study was terminated on November 12, 2024.
Sponsor: Capital Medical University (Other)
Collaborators: China-Japan Friendship Hospital (Other); Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jianping Jia, Director and Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WLB-2022
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active group (Experimental): Take 2 tablets each time (study drug), 3 times a day, a total of 0.9g per day. Take it with warm water half an hour before meals.
  Specifications: 0.15g/ pill (42mg sodium ferulate dihydrate, 42mg rhamnose monohydrate, 66mg chrysin)
  Interventions: Drug: Wei Li Bai capsules
- control group (Placebo Comparator): Take 2 tablets of the control drug (placebo) each time, 3 times a day, 0.9g a day. Take it with warm water half an hour before meals.
  Specification: 0.15g/ grain (microcrystalline cellulose)
  Interventions: Drug: Placebo Comparator of Wei Li Bai capsules

INTERVENTIONS:
Drug: Wei Li Bai capsules — The distribution ratio between the groups was 1:1, and the stratification factor was the degree of illness CDR score. In the study, the entry of each subject into the active group or placebo group will be determined by the randomized system.
  Arms: active group
Drug: Placebo Comparator of Wei Li Bai capsules — The distribution ratio between the groups was 1:1, and the stratification factor was the degree of illness CDR score. In the study, the entry of each subject into the active group or placebo group will be determined by the randomized system.
  Arms: control group

SUMMARY:
In clinical trials of preclinical pharmacodynamic studies, Wei Li Bai capsules has been proved to significantly improve the learning and memory ability of Alzheimer's disease model. In this study, the researchers will use a multicenter, randomized, double-blind, placebo-controlled parallel method to recruit Alzheimer's disease patients to confirm the efficacy and safety of Wei Li Bai capsules. Confirmation of drug efficacy will be observed through changes in Alzheimer's disease patients' general cognitive function scores, scores of different cognitive domains, daily living activities, and symptom severities.

DETAILED DESCRIPTION:
Wei Li Bai Capsule is composed of sodium ferulate tablets, L-rhamnose and chrysin. Sodium ferulate tablet is a domestically marketed drug, L-rhamnose is a marketed food additive, and chrysin is a dietary supplement. All of them have been widely used and their safety has been confirmed. In addition, since these three compounds all show good potential in the treatment of Alzheimer's disease, and play an important role in regulating metabolism, improving blood circulation and anti-inflammatory and antioxidant, this study will explore the synergistic effect of Wei Libai capsule in patients with mild and moderate Alzheimer's disease in 130 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 to 80 years old (including 50 and 80 years old), male or female;
2. Meet the diagnostic criteria of "likely ad dementia" of the National Institute on aging Alzheimer's disease association (NIA-AA) (2011);
3. The subjects are primary school graduates / graduates and above, and have the ability to complete the cognitive ability test and other tests specified in the program;
4. Memory loss lasted for at least 6 months and tended to worsen gradually;
5. Subjects with mild or moderate illness: 11 ≤ total score of MMSE ≤ 26;
6. Total score of Clinical Dementia Rating Scale (CDR):

   Mild dementia: CDR = 1.0; Moderate dementia: CDR = 2.0;
7. The total score of HIS ≤ 4;
8. The total score of Hamilton Depression Scale (HAMD 17 item version) is ≤ 10;
9. If the subject is currently receiving an approved AD treatment, such as acetylcholinesterase inhibitors (AChEI) and/or memantine, they must have been using a stable dose for at least 4 weeks prior to baseline and maintain a stable dose throughout the study;
10. There was no obvious positive sign in nervous system examination;
11. Coronal scanning of head MRI in screening stage: the MTA grade of medial temporal lobe atrophy visual assessment scale is grade 1-2. If the subject can provide the head MRI film that meets the requirements within 3 month before screening, it can be used as the basis for enrollment without repeated shooting; If the researcher cannot judge whether the subject's condition has changed, the coronal MRI scan of the head before enrollment can be added;
12. The subjects should have stable and reliable caregivers, who will take care of them at least 3 days a week and at least 4 hours a day. The caregivers will accompany the subjects to participate in the whole process of the study. Caregivers must accompany the subjects to the study visit and assist the investigator in completing the Neuropsychiatric Inventory (NPI), Alzheimer's Disease Collaborative Study-Ability of Daily Living Scale (ADCS-ADL), and Clinician Interview Based Impression of Severity (CIBIC -plus), and other scale scores;
13. Agree to participate and sign the informed consent form by the legal guardian. Due to the subject's limited cognitive ability and other reasons, the subject's signature is allowed to be left blank, and the reason is explained. In addition, the legal guardian shall sign the reason statement, and the legal guardian shall sign the informed consent.

Exclusion Criteria:

1. During screening, MRI examination showed significant focal lesions, fulfilling one of the following conditions:

   ① There were more than 2 infarcts with diameter > 2 cm at any site;

   ② MRI examination showed that there were infarcts with arbitrary diameter in key parts (such as thalamus, hippocampus, entorhinal cortex, paraolfactory cortex, angular gyrus, cortex and other subcortical gray matter nuclei);

   ③ Fazekas scale grade of white matter lesions >2;

   ④ There are other imaging evidences that do not support mild and moderate AD.
2. Dementia caused by other reasons: vascular dementia, central nervous system infection, Creutzfeldt Jakob disease, Huntington's disease, Parkinson's disease, Lewy body dementia, traumatic dementia, other physical and chemical factors (such as drug poisoning, alcoholism, carbon monoxide poisoning, etc.), important physical diseases (such as hepatic encephalopathy, pulmonary encephalopathy, etc.), intracranial space occupying lesions (such as subdural hematoma, brain tumor), endocrine disorders (such as thyroid disease, parathyroid disease), and vitamin B12, folic acid deficiency or any other known cause;
3. Have suffered from central nervous system diseases (including stroke, optic neuromyelitis, epilepsy, etc.);
4. Subjects who were diagnosed with psychiatric disorders according to DSM-V criteria, including schizophrenia or other mental diseases, bipolar disorder, severe depression or delirium;
5. Abnormal laboratory indexes: liver function (ALT and AST) exceeded 1.5×ULN, renal function (CR) exceeded 1.5×ULN, and creatine kinase exceeded 2×ULN;
6. Untreated hypertensive and hypotensive subjects at screening, or hypertensive subjects with uncontrolled hypertension after treatment; subjects with good blood pressure control after treatment can be determined by the investigator to be suitable for inclusion in this study;
7. Within 1 month of the screening visit, the subject has new or ongoing unstable or serious heart, lung, liver, kidney and hematopoietic diseases according to the judgment of the researcher, and does not meet the conditions for clinical research;
8. Clinically, people with significant allergic reaction history, especially drug allergy history, or known allergy to this product and its excipients;
9. Dyspepsia, esophageal reflux, gastric bleeding or peptic ulcer disease, frequent heartburn (≥ once a week) or any surgical operation that may affect drug absorption (such as partial / total gastrectomy, partial / total small bowel resection and cholecystectomy) within 6 months before screening;
10. Alcohol or drug abusers;
11. Human immunodeficiency virus antibody (ant HIV) and Treponema pallidum antibody (ant TP) are positive;
12. Those who are currently using monoclonal antibody drugs for Alzheimer's disease (e.g., lecanemab, domanemab, etc.), psychotropic drugs, anti-Parkinson drugs, and opioid analgesics within 1 month before the visit;
13. There are uncorrectable visual and auditory disorders, and the neuropsychological test and scale evaluation cannot be completed;
14. Female subjects with positive pregnancy test or lactation and subjects unable to take effective contraceptive measures or have family planning;
15. Participated in other clinical trials within 3 months before the screening visit;
16. There are other situations that the researcher believes are not suitable to participate in this study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive section(ADAS-cog/11) | Change from baseline in ADAS-cog scores at Week 26.
  Differences between the active group in changes in ADAS cog/11 scores (relative to baseline) at weeks 13 and 26 were compared with the placebo group.
  The ADAS-cog assesses cognitive function in seven components: word recall, instruction, structural practice, naming, conceptual practice, orientation, and word recognition. The total score ranges from 0 to 70, with lower scores representing milder disease.

SECONDARY OUTCOMES:
Alzheimer's Disease Co-operative Study Activities of Daily Living (ADCS-ADL) | Change from baseline in ADCS-ADL scores at Week 26.
  Differences between the active group in changes in ADCS-ADL scores (relative to baseline) at weeks 13 and 26 were compared with the placebo group.
  The ADCS-ADL scale can reflect the degree of impairment of the subjects' daily life ability, with a total score of 78 points. The higher the score, the better the subjects' living ability.
Clinician Interview Based Impression of Severity (CIBIC-plus) | Change from baseline in CIBIC-plus scores at Week 26.
  Differences between the active group in changes in CIBIC-plus scores (relative to baseline) at weeks 13 and 26 were compared with the placebo group.
  The CIBIC-plus scale is based on interviews with patients and their caregivers by research physicians to ask, record and assess changes in patients' conditions. Outcomes assessed were: Caregiver Meeting-Clinical Impression Change, Subject Meeting-Clinical Impression Change, and Overall Clinical Impression Change.
Neuropsychiatric Inventory (NPI) | Change from baseline in NPI's 12 behavioral domain scores at week 26.
  Differences in changes in 12-item behavioral domain scores (relative to baseline) on the NPI scale at weeks 13 and 26 between the active group compared with placebo group.
  The NPI scale is an interview conducted by the research doctor based on the patient's caregiver to ask the patient's mental and emotional changes. The questions included 12 items including delusions, hallucinations, depression, and anxiety, each of which identified the severity, frequency, and psychological stress of the caregiver.
Neuropsychiatric Inventory (NPI) | Change from baseline in Caregiver Stress Score on the NPI Scale at Week 26.
  Differences in changes in caregiver stress scores (relative to baseline) on the NPI scale at weeks 13 and 26 between the active group compared with placebo.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - China-Japan Friendship Hospital, Chaoyang, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Xuanwu Hospital of Capital Medical University, Beijing